CLINICAL TRIAL: NCT05216419
Title: Study for Effectiveness in Prevention of Postoperative Hypocalcemia of Preoperative Oral Supplementation of Vitamin D (D-mac 30,000 IU) in Patients Undergoing Total Thyroidectomy
Brief Title: Prevention of Postoperative Hypocalcemia of Oral Vitamin D Supplementation Before Total Thyroidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dalim BioTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Su-jin Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2103-050-1203
Record Dates: First submitted 2021-05-10; First posted 2022-01-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Total Thyroidectomy; Hypocalcemia; Vitamin D Deficiency
MeSH Terms: conditions — Hypocalcemia; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Since the concentration of "D-mac 30,000 IU" in the body reaches the maximum in the body around 1 to 3 weeks after administration, the drug is taken once 15 days before the surgery so that the vitamin D3 concentration is maximized at the time of surgery.
  In the case of the control group, there is no drug to be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Experimental): One dose of "30,000 IU of D-mac" is taken once 15 days prior to surgery.
  Interventions: Drug: Cholecalciferol
- control group (No Intervention): There is no "30,000 IU of D-mac" to be taken.

INTERVENTIONS:
Drug: Cholecalciferol — Since the concentration of "D-mac 30,000 IU" in the body reaches the maximum in the body around 1 to 3 weeks after administration, the drug is taken once 15 days before the surgery so that the vitamin D3 concentration is maximized at the time of surgery.
  In the case of the control group, there is no drug to be taken.
  Arms: case group

SUMMARY:
The hypocalcemia after total thyroidectomy is one of common surgical complications. It may be asymptomatic, but patients can complain of dysfunction around the mouth or extremities, stiffness or convulsion in severe cases. The incidence of transient hypocalcemia was 6.9-46%, and permanent hypocalcemia was reported to be 0.4-33%. It has been reported that the incidence of hypocalcemia after thyroidectomy is high when the difference in blood levels of parathyroid hormone and vitamin D is large before and after surgery.

Therefore, it is a very important task to study the effect of using vitamin D3 (cholecalciferol), which has a better effect on the human body, on the prevention of hypocalcemia after total thyroidectomy with a long follow-up period after surgery. The department of surgery in Seoul National University Hospital intends to analyze the preventive effect "D-mac 30,000 IU" on postoperative hypocalcemia and safety of 'D-mac 30,000 IU" through a prospective randomized clinical trial.

The incidence of postoperative hypocalcemia of the group taking orally taking vitamin D3 (cholecalciferol) before surgery will be compared with that of the group not taking vitamin D3 before surgery. Patients who are enrolled in this RCT are allocated to the case group and the control group. Patients in the case group are taking 30,000 IU of vitamin D3 (cholecalciferol) orally, and patients in the control group are not taking any drugs.

Primary endpoint of this study is to evaluate the incidence of hypocalcemia. And secondary endpoints are to evaluate the recovery duration from postoperative hypocalcemia and the risk factors for postoperative hypocalcemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 70 years old
* Patients undergoing total thyroidectomy due to thyroid disease
* Patients who consented to the study and obtained consent for the study

Exclusion Criteria:

* Patients with confirmed hypocalcemia or hypercalcemia before surgery
* Patients receiving calcium or vitamin D treatment before surgery, patients with excessive vitamin D
* Patients with a previous history of parathyroid disease or a history of cervical irradiation
* Patients with confirmed parathyroid comorbidity
* Patients with diseases or conditions that cause hypercalcemia or hypercalciuria (myeloma, bone metastases, or other malignant bone diseases)
* Patients with confirmed renal dysfunction (glomerular filtration rate <60mL/min/1.73m2) before surgery or with a history of chronic renal failure
* Renal stone disease patient, kidney stone disease patient
* Patients with bowel disease that may affect serum vitamin D levels (celiac disease, small intestine resorption disease, small bowel resection history)
* Patients taking drugs that may affect serum calcium or vitamin D levels (anticonvulsants, bisphosphonates, cisplatin, aminoglycosides, diuretics, proton pump inhibitors, glucocorticoid benzodiazepine derivatives, etc.)
* Uncontrolled hypertension, diabetes, and clotting disorders
* Cardiovascular disease (angina pectoris, heart failure, myocardial infarction, coronary artery disease, history of arrhythmia treatment, stroke, transient ischemic attack), and taking medications for arrhythmia
* Drug Abuse and Alcohol Abuse
* Patients who participated in other drug clinical trials within 30 days
* Patients with a history of allergies to drugs
* For women, pregnant and lactating patients
* Patients judged unsuitable by the person in charge of the clinical trial
* Patients with genetic problems such as galactose intolerance, lactose deficiency, or glucose-galactose malabsorption disorder

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Postoperative hypocalcemia | postoperative 1 day
  The incidence of hypocalcemia at postoperative 1 day
Postoperative hypocalcemia | postoperative 2 weeks
  The incidence of hypocalcemia at postoperative 2 weeks
Postoperative hypocalcemia | postoperative 3 months
  The incidence of hypocalcemia at postoperative 3 months
Postoperative hypocalcemia | postoperative 6 months
  The incidence of hypocalcemia at postoperative 6 months

SECONDARY OUTCOMES:
The occurrence of hypocalcemia sign | 1 day, 2 weeks, 3 months, 6 months after surgery
  The results of survey about the occurrence of hypocalcemia sign
Duration of recovery period from postoperative hypocalcemia | 1 day, 2 weeks, 3 months, 6 months after surgery
  Duration for recovery from hypocalcemia after thyroidectomy
Risk factors for developing postoperative hypocalcemia | 1 day, 2 weeks, 3 months, 6 months after surgery
  Risk factors associated with postoperative hypocalcemia

CONTACTS AND LOCATIONS:
Overall Officials: Su-Jin Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Chung-Ang University Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bahn Chair RS, Burch HB, Cooper DS, Garber JR, Greenlee MC, Klein I, Laurberg P, McDougall IR, Montori VM, Rivkees SA, Ross DS, Sosa JA, Stan MN; American Thyroid Association; American Association of Clinical Endocrinologists. Hyperthyroidism and other causes of thyrotoxicosis: management guidelines of the American Thyroid Association and American Association of Clinical Endocrinologists. Thyroid. 2011 Jun;21(6):593-646. doi: 10.1089/thy.2010.0417. Epub 2011 Apr 21. PMID 21510801
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Ozbas S, Kocak S, Aydintug S, Cakmak A, Demirkiran MA, Wishart GC. Comparison of the complications of subtotal, near total and total thyroidectomy in the surgical management of multinodular goitre. Endocr J. 2005 Apr;52(2):199-205. doi: 10.1507/endocrj.52.199. PMID 15863948
- [Background] Edafe O, Antakia R, Laskar N, Uttley L, Balasubramanian SP. Systematic review and meta-analysis of predictors of post-thyroidectomy hypocalcaemia. Br J Surg. 2014 Mar;101(4):307-20. doi: 10.1002/bjs.9384. Epub 2014 Jan 9. PMID 24402815
- [Background] Alshahrani F, Aljohani N. Vitamin D: deficiency, sufficiency and toxicity. Nutrients. 2013 Sep 13;5(9):3605-16. doi: 10.3390/nu5093605. PMID 24067388
- [Result] Lee GH, Ku YH, Kim HI, Lee MC, Kim MJ. Vitamin D level is not a predictor of hypocalcemia after total thyroidectomy. Langenbecks Arch Surg. 2015 Jul;400(5):617-22. doi: 10.1007/s00423-015-1311-1. Epub 2015 Jun 9. PMID 26050997
- [Result] Thomusch O, Machens A, Sekulla C, Ukkat J, Brauckhoff M, Dralle H. The impact of surgical technique on postoperative hypoparathyroidism in bilateral thyroid surgery: a multivariate analysis of 5846 consecutive patients. Surgery. 2003 Feb;133(2):180-5. doi: 10.1067/msy.2003.61. PMID 12605179
- [Result] Khan Bhettani M, Rehman M, Ahmed M, Altaf HN, Choudry UK, Khan KH. Role of pre-operative vitamin D supplementation to reduce post-thyroidectomy hypocalcemia; Cohort study. Int J Surg. 2019 Nov;71:85-90. doi: 10.1016/j.ijsu.2019.08.035. Epub 2019 Sep 5. PMID 31494332
- [Result] Malik MZ, Mirza AA, Farooqi SA, Chaudhary NA, Waqar M, Bhatti HW. Role of Preoperative Administration of Vitamin D and Calcium in Postoperative Transient Hypocalcemia after Total Thyroidectomy. Cureus. 2019 Apr 30;11(4):e4579. doi: 10.7759/cureus.4579. PMID 31281762